CLINICAL TRIAL: NCT05021406
Title: Extension Study of Carvedilol for the Prevention of the Esophageal Varices Progression on HBV Cirrhotic Patients With Anti-Viral Therapy
Brief Title: Extension Study of Carvedilol RCT Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Xiaojuan Ou, Beijing Friendship Hospital, Beijing Friendship Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-P2-104-04
Record Dates: First submitted 2021-04-18; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-05

CONDITIONS: Liver Cirrhosis; Portal Hypertension
Keywords: Portal Hypertension; Esophageal Varices; Carvedilol
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Esophageal and Gastric Varices | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol+ NUCs therapy (Experimental): Patients randomized to Carvedilol combined with NUCs group during the previous 2-year treatment of RCT study; Patients showed the progression of esophageal varices in NUCs group during the 2-year treatment of RCT study. Based on nucleoside analogue (NUCs), carvedilol will be added to the patients. Carvedilol is started at a dose of 6.25 mg once per day, and will increase to a dose of 12.5 mg once per day after 1 week. Target dose will be maintained at 12.5 mg once per day if patients with systolic blood pressure not lower than 90 mm Hg and HR no less than 50 beats/min.
  Interventions: Drug: Carvedilol 12.5 MG
- NUCs therapy (No Intervention): Continuing take single or combined nucleoside analogue (NUCs) including lamivudine (LAM), adefovir dipivoxil (ADV), entecavir (ETV), telbivudine (TBV), tenofovir disoproxil fumarate (TDF) and tenofovir alafenamide (TAF).

INTERVENTIONS:
Drug: Carvedilol 12.5 MG — Carvedilol is started at a dose of 6.25 mg once per day, and will increase to a dose of 12.5 mg once per day after 1 week. Target dose will be maintained at 12.5 mg once per day if patients with systolic blood pressure not lower than 90 mm Hg and HR no less than 50 beats/min.
  Other Names: Nucleos(t)ide Analogues
  Arms: Carvedilol+ NUCs therapy

SUMMARY:
Patients who have completed 2-years treatment in RCT Study of carvedilol will receive another 2-years extension therapy, aiming to investigate the long-term efficacy of carvedilol for the prevention of esophageal varices in treated HBV cirrhotic patients.

DETAILED DESCRIPTION:
Carvedilol has been shown to be more potent in decreasing portal hypertension than propranolol. But the efficacy of carvedilol to prevent esophageal varices progression in nucleoside analogue (NUCs) treatment HBV related cirrhotic patients was unclear. Previous RCT study aimed to explore the effects of carvedilol for the prevention of the esophageal varices progression on HBV cirrhotic patients with anti-viral therapy has been conducted (NCT03736265). Patients who have completed 2-years treatment in RCT Study of carvedilol will receive another 2-years extension therapy, aiming to investigate the long-term efficacy of carvedilol for the prevention of esophageal varices in treated HBV cirrhotic patients. Patients were allocated according to the outcome of EDGs at 2-year during RCT study. Patients will be assessed at baseline and every six months for blood cell count, liver function test, HBVDNA, AFP, prothrombin time, liver ultrasonography, and Fibroscan. A third EGDs will be performed at 4-year.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed the 2-year RCT study of carvedilol in HBV cirrhotic patients with anti-viral therapy;
* Subjects who are willing to participate the extension study.

Exclusion Criteria:

* Subjects who refused to receive 2-year EGD examination during the previous RCT study;
* Subjects who could not compliance with the protocol judged by investigators;
* Subjects who are not suitable for the study judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
The progression incidence of esophageal varices after 4-year therapy | 4-year
  Progression of esophageal varices defines as follows:
  1. Varices developed from small (F1) to medium or large (F2/F3)
  2. Varices developed from medium (F2) to large (F3)
  3. New-onset red sign without change in the degree of varices.
  4. Bleeding from esophageal varices.

SECONDARY OUTCOMES:
The incidence of liver cirrhosis decompensation | 4-year
  Cumulative rate of liver cirrhosis decompensation, including bleeding, ascites, hepatic encephalopathy, ect.
The incidence of hepatic cellular carcinoma, death or liver transplantation. | 4-year
  Cumulative rate of hepatic cellular carcinoma, death or liver transplantation.
The change of non-invasive assessment score reflecting liver fibrosis. | 4-year
  Higher scores mean a worse outcome.
The change of non-invasive assessment score reflecting liver function. | 4-year
  Higher scores mean a worse outcome.
The dynamic change of liver stiffness quantified by transient elastography. | 4-year
  The dynamic change of liver stiffness quantified by transient elastography.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojuan Ou, Principal Investigator — Beijing Friendship Hospital
Locations (14):
- China (14):
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Affiliated Hospital of Yanbian University, Yanji, Jilin
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality
  - Tianjin Third Central Hospital, Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Xiqing Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Uygur Autonomous Region Traditional Chinese Medicine Hospital, Xinjiang, Xinjiang

IPD SHARING:
Plan to Share IPD: No